CLINICAL TRIAL: NCT05972239
Title: Balance Training: Its Effect on Pulmonary Rehabilitation of Elderly Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Balance Training in Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Elisabetta Zampogna, Dr, Istituti Clinici Scientifici Maugeri SpA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2763
Record Dates: First submitted 2023-05-23; First posted 2023-08-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: COPD
Keywords: Exercise; Rehabilitation; Aged; postural balance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Educational interventions, aerobic and strenght training, flexibility exercises.
  Interventions: Other: Standard pulmonary rehabilitation program
- Intervention (Experimental): Educational interventions, aerobic and strenght training, balance training.
  Interventions: Other: Balance training added on standard pulmonary rehabilitation

INTERVENTIONS:
Other: Standard pulmonary rehabilitation program — Educational interventions, 3 individual sessions of 10-20 minutes and 1 weekly group meeting of 45-60 minutes on nutrition and on the emotional management of the disease. Supervised and incremental aerobic training, lasting at least 30 minutes, 5/6 days a week for a total of 12-14 sessions. The initial workload will be set between 50-70% of the maximum load (watts) determined starting from the 6MWT using the Hill equation and will be increased to reach a perception of moderate-intense fatigue and/or dyspnea. Supervised strength training of the lower limbs and upper limbs, lasting 30 minutes, 5/6 times a week for a total of 12-14 sessions. The workload will be calibrated to allow the execution of 12 consecutive repetitions and will be progressively increased by 0.5 kg in order to cause a moderate/intense fatigue and/or dyspnea. Group exercises aimed at improving flexibility of the trunk, lower and upper limbs, lasting at least 30 minutes, 5/6 days a week, for a total of 12-14 sessions.
  Arms: Control
Other: Balance training added on standard pulmonary rehabilitation — Educational interventions, 3 individual sessions of 10-20 minutes and 1 weekly group meeting of 45-60 minutes on nutrition and on the emotional management of the disease. Supervised and incremental aerobic training, lasting at least 30 minutes, 5/6 days a week for a total of 12-14 sessions. The initial workload will be set between 50-70% of the maximum load determined from the 6MWT (Hill equation) and will be increased based on dyspnea. Supervised strength training of the lower limbs and upper limbs, lasting 30 minutes, 5/6 times a week for a total of 12-14 sessions. The workload will be progressively increased. Supervised balance training sessions lasting 30 minutes, 5/6 times a week for a total of 12-14 sessions. The sequence of the exercises will be personalized according to the result of the Berg Balance Scale and modified according to the progress.
  Arms: Intervention

SUMMARY:
The aim of the study will be to verify whether the addition of an exercise program aimed to improve balance can reduce the risk of falling in subjects with COPD over 80 years of age compared to the standard rehabilitation program. Patients will be randomly assigned in two groups (intervention and control). The pulmonary rehabilitation (PR) program is organized in accordance with current guidelines.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease-COPD is the most prevalent pathology among chronic airway diseases. The average age of life has increased. Subjects over 80 years old have peculiar characteristics. Individuals with COPD have an increased risk of falling compared with healthy peers. A pulmonary rehabilitation program reduces the risk of falling as measured by gait speed. Balance training on the elderly has been shown to be effective in improving muscle strength, coordination, balance and in reducing the risk and number of falls and the fear of falling.

The enrolled subjects will complete an in-patient PR program according to enrollment.

Control: education, aerobic and strength training and callisthenic exercises. Intervention: education, aerobic and strength training as group Control and balance training. At baseline will be recorded: demographics and anthropometrics, comorbidities, drug therapy, flow/volume curve, arterial blood gases, serum hemoglobin, history of fall, exacerbations and risk of sarcopenia. Before and after the PR the following outcome measures will be assessed: balance performance, peripheral muscle strength, gait speed, health status, dyspnea, quality of life, exercise capacity, confidence with balance and perceived change. Sample size calculation was performed based on the primary endpoint of the study. We estimate a number of 50 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years old,
* Diagnosis of COPD according to GOLD Guidelines (Tiffenau Index <70%) under optimized medical treatment,
* Able to perform and complete study procedures.

Exclusion Criteria:

* Anticholinergic Cognitive Burden score ≥3,
* Mini-Mental State Examination <22,
* Acute or chronic impairment and/or medical diseases that are likely to preclude exercise testing and PR.
* Brain lesions,
* Inner ear disease
* Visual deficit,
* Lower limb surgery in the previous 6 months.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 3 weeks
  Berg Balance Scale (BBS). Scores range from 0 (worst) - 4 (best).

SECONDARY OUTCOMES:
Peripheral muscle strenght | 3 weeks
  Five sit to stand test (5STS). Time < 14.9 seconds (best), >14.8 seconds (worst).
Gait speed | 3 weeks
  4-meter gait speed test (4MGS). Time < 4.83 seconds (best), >4.82 seconds (worst).
Health status | 3 weeks
  The COPD Assessment Test (CAT) score ranges from 0 (best) to 40 (worst).
Dyspnea | 3 weeks
  Medical Research Council (mMRC) score ranges from 0 (best) to 4 (worst).
Dyspnea on daily life activities | 3 weeks
  Barthel Dyspnea Index (BDI) total score ranges from 0 (best) to 100 (worst).
COPD Quality of life | 3 weeks
  EuroQoL-5D total score ranges from 0 (worst) to 100 (best).
Exercise capacity | 3 weeks
  Six-Minute Walking Test (6MWT) measures the maximum walked distance in meters (m) in a given time (6 minutes).
Confidence with balance | 3 weeks
  Activities-specific Balance Confidence short form (ABC-6) Scale. Score from 0 (worst) to 100 (best).
Perceived change | 3 weeks
  Global perceived effect (GPE) scale. Score range from 1 (best) to 7 (worst).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of pulmonary rehabilitation, Tradate, Varese, Italy

IPD SHARING:
Plan to Share IPD: No